CLINICAL TRIAL: NCT06418438
Title: To Compare the Clinical Efficacy and Safety of Laparoscopic Uterosacral Ligament Suspension With or Without Hysterectomy in the Treatment of POP
Brief Title: A Randomized Controlled Trail of Uterosacral Ligament Suspension in the Treatment of Pelvic Organ Prolapse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lan Zhu (Other)
Responsible Party: Sponsor-Investigator, Lan Zhu, Director of the Department of Obstetrics and Gynecology at Peking Union Medical College Hospital, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K5787
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic uterosacral ligament suspension with hysterectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic uterosacral ligament suspension with hysterectomy
- Laparoscopic uterosacral ligament suspension with cervical amputation (Experimental)
  Interventions: Procedure: Laparoscopic uterosacral ligament suspension with cervical amputation

INTERVENTIONS:
Procedure: Laparoscopic uterosacral ligament suspension with hysterectomy — After anesthesia, bladder stone removal patients undergo laparoscopic hysterectomy. The adnexa are coagulated and cut, and the bladder peritoneal reflection is opened. The uterus is removed transvaginally. Next, laparoscopic uterosacral ligament suspension is performed. The right and left uterosacral ligaments are freed and sutured to lift the residual end.
  Arms: Laparoscopic uterosacral ligament suspension with hysterectomy
Procedure: Laparoscopic uterosacral ligament suspension with cervical amputation — After anesthesia, bladder stone removal patients undergo cervical amputation surgery. The cervix is exposed and elevated using Allis forceps. A dilator is used to expand the cervix, and an incision is made on the anterior vaginal wall. The cervix is excised and shaped using the Sturmdorf method. Afterward, laparoscopic uterosacral ligament suspension is performed. The right and left uterosacral ligaments are freed and sutured to lift the uterus.
  Arms: Laparoscopic uterosacral ligament suspension with cervical amputation

SUMMARY:
Pelvic organ prolapse (POP) is one of the common benign gynecological disorders in middle-aged and elderly women, which severely affects patients' quality of life and increases the social burden. The lifetime risk of undergoing surgery for POP is 12.6%. Surgery is an important treatment modality for POP, and currently, there are various surgical procedures used in clinical practice, but there is still no clear consensus on which procedure is superior. Autologous tissue repair remains crucial in pelvic floor reconstruction surgery, and high uterosacral ligament suspension (HUSLS) via a vaginal approach is a classic corrective procedure for central pelvic defects. However, with the development of minimally invasive techniques, laparoscopic uterosacral ligament suspension (LUSLS) has been widely used in the field of pelvic floor reconstruction. Compared to the vaginal approach, LUSLS is easier to perform, has a shorter learning curve, provides better exposure of the ureters, and allows for higher-quality suture placement under safe conditions. The main controversial clinical issue in the industry regarding high uterosacral ligament suspension is whether to perform uterine preservation, with the core concern being the risk of postoperative recurrence. High uterosacral ligament suspension with uterine preservation achieves level I repair by fixing the lower segment or cervix to supporting structures. Its advantages include shorter operation time, less blood loss, and the preservation of the patient's fertility. Many women request uterine preservation for various reasons. Therefore, high-quality research is needed to guide the clinical decision-making regarding uterine preservation in high uterosacral ligament suspension. Previous studies have found that approximately 40% of patients with pelvic organ prolapse have concurrent cervical elongation. For patients with cervical elongation, symptoms in the central pelvic region are mainly caused by the protrusion of elongated cervical tissue into the vagina. Removing the elongated cervix significantly reduces the need for biological support in pelvic floor reconstruction, making autologous tissue repair strategies the preferred option for this patient population while providing a foundation for uterine preservation. Based on long-term observational studies, the Department of Obstetrics and Gynecology at Peking Union Medical College Hospital has proposed combining laparoscopic uterosacral ligament suspension with cervical amputation for the treatment of pelvic organ prolapse with cervical elongation. This study aims to compare whether uterine preservation in laparoscopic uterosacral ligament suspension is non-inferior to uterine removal, providing more treatment options for future patients with pelvic organ prolapse and cervical elongation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with symptomatic stage II or higher uterine prolapse (C ≥ +1cm) and gynecological ultrasonography confirming cervical length ≥ 4cm. Concurrent anterior and/or posterior vaginal wall prolapse may be present.
* Preoperative pelvic ultrasound and cervical screening show no abnormalities.
* The patient does not have a desire for future fertility.
* Willingness and ability to adhere to the follow-up treatment plan.
* Competence to provide informed consent.

Exclusion Criteria:

* Suspected untreated lower genital tract tumor, accompanied by other uterine, ovarian, and cervical lesions requiring surgical intervention, indicating contraindication for uterine preservation.
* Patients with a history of total hysterectomy/subtotal hysterectomy.
* Patients who have previously undergone pelvic organ prolapse surgery or other pelvic floor surgeries.
* Patients with contraindications for laparoscopic surgery, such as intestinal obstruction.
* Patients with intestinal hernia.
* Patients with gynecological and urinary tract infections, anticoagulant therapy, coagulation disorders, previous pelvic radiotherapy, as well as neurological or medical conditions affecting bladder and bowel function (such as multiple sclerosis, spinal cord injury, or residual neurological dysfunction caused by stroke), and patients with underlying conditions such as chronic pelvic pain, who are at higher risk for surgery.
* Simultaneous anti-urinary incontinence surgery is required for this procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The composite success rate at the one-year follow-up | At the one-year follow-up
  1. No sensation of vaginal bulge or protrusion, indicated by a response of "no" or a score of 0 on question 3 of the PFDI-20 questionnaire, which asks, "Do you often see or feel a bulge or something falling out of your vagina?"
  2. No further treatment (surgical or non-surgical) required for POP (Pelvic Organ Prolapse).
  3. Absence of POP-Q points at the hymen or beyond the hymen, indicating that Aa, Ba, C, Ap, and Bp are all < 0cm.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No